CLINICAL TRIAL: NCT01849445
Title: Targeted Rehabilitation to Improve Outcome After Knee Replacement- A Physiotherapy Study (TRIO-Physio)
Brief Title: Targeted Rehabilitation to Improve Outcome After Knee Replacement- A Physiotherapy Study
Acronym: TRIO-Physio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arthritis Research UK 20100; 13\SS\0051 (Other: South East Scotland REC 01)
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive physiotherapy (Active Comparator): Participants will visit hospital for physiotherapy sessions once a week for 6 weeks in addition to completing prescribed exercises twice a week at home on their own.
  Interventions: Procedure: Intensive physiotherapy
- Home physiotherapy excercises (Active Comparator): Patients will be asked to complete prescribed exercises at home on their own 3 times a week for 6 weeks.
  Interventions: Other: Home physiotherapy exercises

INTERVENTIONS:
Procedure: Intensive physiotherapy — Participants will visit hospital for physiotherapy sessions once a week for 6 weeks in addition to completing prescribed exercises twice a week at home on their own.
  Arms: Intensive physiotherapy
Other: Home physiotherapy exercises — Patients will be asked to complete prescribed exercises at home on their own 3 times a week for 6 weeks.
  Arms: Home physiotherapy excercises

SUMMARY:
The TRIO-physio study is looking at how well patients with osteoarthritis recover after knee replacement surgery (also known as Total Knee Arthroplasty (TKA)). Currently around 20% of patients are not satisfied after TKA. This project will look to find out if the research team can identify patients who will not recover well at an earlier stage, so that these patients can be helped sooner.

The study will try to determine if doing intense physiotherapy with patients who are not doing well at the first review (6 weeks after their operation) can improve how well they have recovered at one year.

DETAILED DESCRIPTION:
The study is a randomised controlled trial comparing the effect of intensive physiotherapy compared to current standard of care therapy, targeted to patients performing poorly at 6 weeks following total knee replacement.

All patients will be made aware of the study pre-operatively at the recruiting centres. Prior to surgery they will complete the routine pre-operative outcome assessment questionnaires (Oxford Knee Score and EQ-5D) as part of the national PROMS program and then undergo the local standard total knee replacement and immediate post-operative care pathway.

All patients will be routinely reviewed 6 weeks post-operatively by the usual clinical teams. At this review the Oxford Knee Score will again be assessed. Those patients who report a score of 26 or less (on the 0-48 OKS scoring system), which is defined as poor by the Kalairajah classification (Kalairajah, 2005), will be approached to consent. If consent is given and the patient is eligible to enter the trial, randomisation into one of the following groups will occur: to standard care (encompassing a one off physiotherapy review, 6 weeks of home exercise prescription and final review) or to an interventional arm, where 18 sessions of structured physiotherapy will be administered over a 6 week period, where 6 of these sessions will be 'contact sessions' performed under the supervision of the physiotherapist.

All trial participants will be reviewed immediately post intervention (i.e. at 14 weeks post operation) and then by postal questionnaire at 26 and 52 weeks post-operation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary total knee arthroplasty for osteoarthritis.
* Defined poor outcome (Oxford Knee Score less than or equal to 26) at first post-op review (6 weeks).
* Patients are able to consent and willing to comply with the study protocol

Exclusion Criteria:

* Patients undergoing revision knee arthroplasty or fully constrained knee arthroplasty
* Knee replacement for a diagnosis other than osteoarthritis
* Patients unable to attend the study physiotherapy intervention centre
* Procedures done purely for pain relief (such as for patients with no walking capacity)
* Patients already receiving ongoing structured post-operative exercise rehabilitation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score | 52 weeks post-operation
  Primary analysis will be 52 week outcome (Oxford Knee Score) in the enhanced physiotherapy intervention group compared to the current standard of care physiotherapy treatment group.

SECONDARY OUTCOMES:
Patient satisfaction | 52 weeks post-operation
  Assess patient satisfaction with knee arthroplasty. Assessed with a specific patient satisfaction question:
  Are you satisfied with your knee replacement? (Possible responses: very satisfied, satisfied, dissatisfied, very dissatisfied) Specific satisfaction with pain relief and functional ability will also be assessed. 4 additional sub-questions relating to facets of satisfaction:
  1. "How well did the surgery relieve the pain in your affected joint?"
  2. "How well did the surgery increase your ability to perform regular activities?"
  3. "How well did the surgery allow you to perform heavy work or sport activities?"
  4. "How well did the surgery meet your expectations?"
  (Possible answers: excellently, very well, well, fairly, poorly)
Knee function | week 8 and week 14
  Assess the actual physical function of the patient as a result of the differing physiotherapy interventions. Timed-get-up-and-go-test, assessed prior to (8-weeks post op) and following 6 week physiotherapy protocol (14 weeks post-op).
Cost effectiveness | 52 weeks post
  To evaluate the cost effectiveness of enhanced targeted physiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hamish Simpson, Principal Investigator — University of Edinburgh
Locations (6):
- United Kingdom (6):
  - NHS Grampian, Aberdeen
  - Doncaster Royal Infirmary, Doncaster
  - NHS Lothian, Edinburgh
  - Oxford University Hospitals NHS Trust, Oxford
  - Kim Brown, Portsmouth
  - Weston Super Mare, Weston-super-Mare

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamilton DF, Beard DJ, Barker KL, Macfarlane GJ, Tuck CE, Stoddart A, Wilton T, Hutchinson JD, Murray GD, Simpson AHRW; TRIO investigators. Targeting rehabilitation to improve outcomes after total knee arthroplasty in patients at risk of poor outcomes: randomised controlled trial. BMJ. 2020 Oct 13;371:m3576. doi: 10.1136/bmj.m3576. PMID 33051212
- [Derived] Simpson AH, Hamilton DF, Beard DJ, Barker KL, Wilton T, Hutchison JD, Tuck C, Stoddard A, Macfarlane GJ, Murray GD. Targeted rehabilitation to improve outcome after total knee replacement (TRIO): study protocol for a randomised controlled trial. Trials. 2014 Feb 1;15:44. doi: 10.1186/1745-6215-15-44. PMID 24484541